CLINICAL TRIAL: NCT04955925
Title: Comparison of the Effect of Sevoflurane and Propofol on the Optic Nerve Sheath Diameter in Patients Undergoing Middle Ear Surgery
Brief Title: Effect of Sevoflurane and Propofol on the Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 03-2020
Record Dates: First submitted 2021-03-31; First posted 2021-07-09 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Optic Nerve Sheath Diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sevoflurane group: Anesthesia is maintained with sevoflurane during the surgery.
  Interventions: Diagnostic Test: Ultrasound examination of the optic nerve sheath diameter
- Propofol group: Anesthesia is maintained with total venous anesthesia using propofol during the surgery.
  Interventions: Diagnostic Test: Ultrasound examination of the optic nerve sheath diameter

INTERVENTIONS:
Diagnostic Test: Ultrasound examination of the optic nerve sheath diameter — The optic nerve sheath diameter is examined using ultrasonography.

SUMMARY:
In the present study, we compare the effect of sevoflurane and propofol on the optic nerve sheath diameter in patients undergoing middle ear surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing middle ear surgery

Exclusion Criteria:

* History of cerebrovascular diseases
* Increased intracranial pressure
* History of ophthalmic surgery or diseases

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing middle ear surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Change of the optic nerve sheath diameter | At 1 minute after the induction of anesthesia and at 1 minute after the end of surgery
  The optic nerve sheath of each eye is observed using ultrasound, and the optic nerve sheath diameter is assessed after induction of anesthesia and at the end of surgery.

SECONDARY OUTCOMES:
Optic nerve sheath diameter at each time point | At 1 minute after the induction of anesthesia and at 1 minute after the end of surgery
  The optic nerve sheath of each eye is observed using ultrasound, and the optic nerve sheath diameter is assessed after induction of anesthesia and at the end of surgery.
Nausea and vomiting | At 1 hour after surgery
  Presence and severity of nausea and vomiting is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea